CLINICAL TRIAL: NCT06528431
Title: Design and Evaluation of an Individualized Biodrug Tapering Strategy Based on Biodrug Dosage: the MONITORA Study
Acronym: MONITORA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: AAP MESSIDOR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24CH046; 2024-514313-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Adalimumab; Remission management; step wedge trial
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Randomization comparing 2 therapeutic strategies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single arm trial (Experimental): Single arm trial in patients with established RA who achieved clinical remission with subcutaneous injection of adalimumab in combination with MTX (methotrexate). Patients will undergo a tapering strategy based only on the clinical status (flare /no flare) during 12 months.
  Interventions: Drug: Clinical tapering strategy
- Maintenance arm (No Intervention): Maintenance arm: the same adalimumab regimen
- Optimized tapering adalimumab (Experimental): An optimized tapering adalimumab strategy based on the disease activity and the adalimumab trough concentration. The tapering strategy will rely on the adalimumab trough concentration. Spacing will be performed only if adalimumab trough concentration is above the pre-specified concentration threshold
  Interventions: Drug: Step Wedge trial

INTERVENTIONS:
Drug: Clinical tapering strategy — Clinical Tapering strategy : Adalimumab injections will be progressively spaced out according to DAS28 assessment every 3 months
  Arms: Single arm trial
Drug: Step Wedge trial — Step Wedge trial : At baseline, all the patients will receive in this study the standard adalimumab dosing regimen. At subsequent time points (steps), patients will begin the intervention of interest, here the tapering adalimumab strategy. The time at which a patient begins the intervention will be randomized. We fixed the time steps duration to 3 months that corresponds the frequency of there commended follow-up of RA patients
  Arms: Optimized tapering adalimumab

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory joint disorder. Since twenty year and the use of synthetic disease-modifying anti-rheumatic drugs (csDMARDs) and biological (b)DMARD, remission can be reached. When remission is obtained, the physician has no recommendations for managing a step-down, and future guidelines will be useful to assist the clinician. Recent data suggest that tapering is feasible, but with high risk of flares. Flares are less frequent when bDMARD blood concentration is high. But, the optimal adalimumab concentration to keep before a step of tapering no targeting personal is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patients with a diagnosis of RA according to ACR/EULAR 2010 criteria
* Remission according to DAS28<=2.6 for at least 6 months
* Patient treated with ADA for at least 6 months. The patient is treated according to one of the following two strategies:
* ADA 40 mg every two weeks (= every 14 days) according to the standard regimen
* or ADA 40 mg every 3 weeks (= every 21 days)
* A negative highly sensitive pregnancy test for women of Childbearing Potential*
* Affiliated person or beneficiary of a social security scheme
* Informed consent signed by the patient after information

Exclusion Criteria:

* Incapacity or refusal to understand and / or sign informed consent to participate in the study.
* Existing pregnancy, lactation, or intended pregnancy within the next 15 months
* Fibromyalgia associated to RA
* Any dose of prednisone for RA treatment 6 months before inclusion
* Patient deprived of liberty or patient under guardianship or curator ship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-09-19 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
Rheumatoid arthritis flare-up | 15 Months
  The RA flare-up will be defined as previously by:
  1. a disease activity score (DAS)28 that increase above 2.6 for patient previously in remission (DAS28≤2.6) and a DAS28 increase (ΔDAS28) of 0.6 or greater for patients with low disease activity (2.6<DAS28<3.2) : YES/NO
  2. Use of a glucocorticoid for the symptoms of RA, regarless of the DAS28 : YES/NO
  DAS28 is calculated according to the formula that is composed of the number of tender joints (TJC) and swollen joints (SJC), patient's global assessment of disease activity on a visual analogue scale (PGA, 0-10), and C-reactive protein (CRP).
  Formula for calculating DAS28 using C-reactive protein (CRP) :
  DAS28-CRP=(0.56 × √TJC) + (0.28 × √SJC) + (0.014 × PGA [mm]) + (0.36 × ln(CRP in mg/L+1) + 0.96,

SECONDARY OUTCOMES:
Infection | 15 months
  Number of infection

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Infirmerie Protestante, Caluire-et-Cuire
  - Chd Vendee, La Roche-sur-Yon
  - Hopital Philibert, Lomme
  - Chu Montpellier, Montpellier
  - Ap-Hp Pitie Salpetriere, Paris
  - Chu Reims, Reims
  - Chu Saint Etienne, Saint-Etienne
  - Chru Tours, Tours